CLINICAL TRIAL: NCT05037019
Title: Single Fraction Preoperative Radiation as a Strategy for Local Control of Breast Cancer During a COVID-19 Pandemic
Brief Title: SIGNAL During a COVID-19 Pandemic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgery wait times during the COVID-19 pandemic were eventually reduced to pre-pandemic wait times. This study became irrelevant.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115858
Record Dates: First submitted 2020-05-05; First posted 2021-09-08 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: radiation therapy; radiotherapy; breast cancer; SBRT; neoadjuvant radiation; hypofractionation; stereotactic; preoperative
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single fraction radiotherapy (Experimental): Single fraction of 21 Gy stereotactic radiation therapy delivered to a single malignant lesion of the breast prior to any other treatment for breast cancer.
  Interventions: Procedure: Radiation therapy

INTERVENTIONS:
Procedure: Radiation therapy — Women diagnosed with early stage breast cancer are given a single dose of stereotactic body radiation therapy (SBRT) prior to any other treatment in the context of delayed lumpectomy due to the COVID-19 pandemic.
  Other Names: Radiotherapy; Stereotactic body radiation therapy (SBRT)

SUMMARY:
The standard treatment for early stage, estrogen-receptor positive breast cancer is lumpectomy and sentinel lymph node biopsy followed by 16-25 treatments of adjuvant whole-breast radiation therapy plus or minus hormone therapy. However, the COVID-19 pandemic has necessitated changes in the way breast cancer is treated in order to reduce contact between individuals, reduce spread of the novel coronavirus, and lessen the impact on health care resources. As elective surgeries are being cancelled, current pandemic guidelines recommend that patients be started on hormone treatment while waiting for surgeries to be re-instated. Only after this surgery occurs will patients receive radiation treatment, dramatically extending the time between diagnosis and end of treatment. Emergency pandemic guidelines in the UK and other countries recommend 5 fractions of pre-operative radiation therapy where appropriate. Based on previous work in the SIGNAL 1.0 and SIGNAL 2.0 clinical trials, the investigators are proposing treating patients with early stage breast cancers with one single fraction of stereotactic neoadjuvant radiation during the pre-operative waiting period. This will allow patients to complete radiation therapy upfront while reducing the number of patient visits to hospital. This will also allow investigators to evaluate the ability of single-fraction targeted radiation to induce a pathologic complete response.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥ 50 years old
* Postmenopausal
* Tumor size < 3cm on pre-treatment imaging
* Any grade of disease, estrogen receptor (ER) positive, HER2 negative
* Unicentric/unifocal disease
* Invasive ductal carcinoma or other favorable subtypes of epithelial breast malignancy (lobular, medullary, papillary, colloid, mucinous, or tubular) .
* Clinically node-negative (based upon pre-treatment physical examination and/or axillary ultrasound).
* Surgical expectation that a > 2mm margin can be obtained.
* Lesion is 1 cm or greater from the skin surface.
* Able to lie comfortably in the prone position with arms raised above the head for extended periods of time.

Exclusion Criteria:

* Male sex
* Under 50 years of age
* Previous RT to the same breast
* HER2 positive disease
* Evidence of suspicious diffuse microcalcifications in the breast prior to the start of radiation.
* Local metastatic spread into ipsilateral axilla and/or supraclavicular region and/or neck nodes and/or internal mammary nodes diagnosed on clinical examination or any imaging assessment (unless such sites can be confirmed as negative following biopsy)
* Distant metastases
* Involvement of contralateral axillary, supraclavicular, infraclavicular or internal mammary nodes (unless there is histologic confirmation that these nodes are negative)
* Prior non-hormonal therapy or radiation therapy for the current breast cancer
* Patients with Paget's disease of the nipple.
* Skin involvement, regardless of tumor size.
* Patients with a breast technically unsatisfactory for radiation therapy.
* Inability to lie prone with arms raised above head for extended periods of time.
* Patients not appropriate for BCS due to expectation of poor cosmetic result, even without RT
* Collagen vascular disease (particularly lupus, scleroderma, dermatomyositis)
* Inability or unwillingness to provide informed consent.
* Any other malignancy at any site (except non-melanomatous skin cancer) < 5 years prior to study enrollment
* Patients who are pregnant or lactating

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 1 year
  To evaluate whether a pathologic complete response can be achieved when radiotherapy is delivered in a single 21 Gy fraction, establishing whether tumour response has a linear function with time in the context of delayed surgery. Pathologic complete response will be treated as a dichotomous variable (yes/no). Results will be stratified based on whether patients were also placed on neoadjuvant hormone treatment.
Feasibility of SBRT during a pandemic | 1 year
  To demonstrate feasibility of treating early stage breast cancer patients with a single 21 Gy fraction during the COVID-19 pandemic. This will be measured by accrual rate and the number of patients that can be treated during this pandemic.

SECONDARY OUTCOMES:
Radiation toxicity | 1.5 years
  A secondary objective is to evaluate toxicity resulting from delivering radiation therapy in this manner. Toxicity will be evaluated using the CTCAE grading system.
Cosmesis | 1.5 years
  A secondary objective is to evaluate breast cosmesis resulting from delivery of radiation therapy in this manner. Cosmesis will be evaluated using the Modified Harvard-Harris Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No